CLINICAL TRIAL: NCT06509789
Title: Optimizing the Intensity of Priming Theta Burst Stimulation to Improve Hemiparetic Upper Limb Motor Functions After Stroke: a Randomized Controlled Trial
Brief Title: Priming Theta Burst Stimulation for Stroke: A Study of Intensity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Tung Wah Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20240229001
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2024-07

CONDITIONS: Stroke
Keywords: Stroke; Transcranial magnetic stimulation; Theta burst stimulation
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation; Clinical Protocols

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low intensity priming intermittent theta burst stimulation (iTBS) (Experimental): Standard 600-pulse TBS will be applied using the MagPro X100 stimulator (MagVenture, Denmark) connected with a figure-of-eight coil (Cooling B-65). The resting motor threshold (RMT) of the motor cortex (M1) will be defined as the minimum intensity over the motor hotspot that could elicit an motor evoked potential (MEP) of no less than 50 μv over the first dorsal interosseous muscle in at least five out of 10 trials. Low intensity priming iTBS consists of a session of 55% RMT cTBS, followed by 70% RMT iTBS.
  Interventions: Device: Transcranial magnetic stimulation (TMS) - Theta burst stimulation (TBS) protocol
- Standard priming intermittent theta burst stimulation (iTBS) (Experimental): Standard 600-pulse TBS will be applied using the MagPro X100 stimulator (MagVenture, Denmark) connected with a figure-of-eight coil (Cooling B-65). The resting motor threshold (RMT) of the motor cortex (M1) will be defined as the minimum intensity over the motor hotspot that could elicit an motor evoked potential (MEP) of no less than 50 μv over the first dorsal interosseous muscle in at least five out of 10 trials. Standard priming iTBS consists of a session of 70% RMT cTBS, followed by 70% RMT iTBS.
  Interventions: Device: Transcranial magnetic stimulation (TMS) - Theta burst stimulation (TBS) protocol
- Nonpriming intermittent theta burst stimulation (iTBS) (Active Comparator): Standard 600-pulse TBS will be applied using the MagPro X100 stimulator (MagVenture, Denmark) connected with a figure-of-eight coil (Cooling B-65). The resting motor threshold (RMT) of the motor cortex (M1) will be defined as the minimum intensity over the motor hotspot that could elicit an motor evoked potential (MEP) of no less than 50 μv over the first dorsal interosseous muscle in at least five out of 10 trials. Nonpriming iTBS consists of a session of 20% RMT cTBS (sham), followed by 70% RMT iTBS.
  Interventions: Device: Transcranial magnetic stimulation (TMS) - Theta burst stimulation (TBS) protocol
- Sham stimulation (Sham Comparator): Standard 600-pulse TBS will be applied using the MagPro X100 stimulator (MagVenture, Denmark) connected with a figure-of-eight coil (Cooling B-65). The resting motor threshold (RMT) of the motor cortex (M1) will be defined as the minimum intensity over the motor hotspot that could elicit an motor evoked potential (MEP) of no less than 50 μv over the first dorsal interosseous muscle in at least five out of 10 trials. Sham stimulation consists of a session of 20% RMT cTBS (sham), followed by 20% RMT iTBS (sham).
  Interventions: Device: Transcranial magnetic stimulation (TMS) - Theta burst stimulation (TBS) protocol

INTERVENTIONS:
Device: Transcranial magnetic stimulation (TMS) - Theta burst stimulation (TBS) protocol — This procedure uses magnetic fields to stimulate nerve cells in the brain involved in various neurological functions, such as motor control. Theta burst stimulation is a patterned form of TMS protocol.

SUMMARY:
Objectives: To compare the effects of low intensity priming intermittent theta burst stimulation (iTBS) with those derived from conventional intensity priming iTBS, nonpriming iTBS, and sham stimulation in terms of improving hemiparetic upper limb motor functionality and modulating cortical excitation/inhibition in patients with stroke.

Hypothesis to be tested: We hypothesize that low intensity priming iTBS can maximize the induction of therapeutically beneficial metaplasticity, and that this will be reflected in enhanced cortical excitation and reduced cortical inhibition, thereby enabling superior upper limb motor recovery in patients with stroke.

Design and subjects: A randomized controlled trial involving 108 patients with chronic stroke.

Study instruments: Transcranial magnetic stimulation (TMS) and electroencephalography (EEG).

Interventions: Participants will be randomly assigned into one of the following four groups: (1) low intensity priming iTBS (55% resting motor threshold [RMT] continuous theta burst stimulation [cTBS]+70% RMT iTBS); (2) conventional intensity priming iTBS (70% RMT cTBS+70% RMT iTBS); (3) nonpriming iTBS (sham cTBS+70% RMT iTBS); and (4) sham stimulation (sham cTBS+sham iTBS). All participants will receive 60-minute standard motor training after completion of the stimulation program. The intervention will last four weeks, with three sessions per week.

Main outcome measures: Upper limb motor tests and levels of cortical excitation/inhibition measured by TMS-evoked EEG potentials.

Data analysis: Analysis of variance (ANOVA). Expected results: The low intensity priming iTBS protocol will be the most efficacious protocol for enhancing cortical excitation and reducing cortical inhibition in post-stroke patients and will thereby produce superior outcomes with regard to upper limb motor functionality.

DETAILED DESCRIPTION:
Objectives: To compare the effects of low intensity priming intermittent theta burst stimulation (iTBS) with those derived from conventional intensity priming iTBS, nonpriming iTBS, and sham stimulation in terms of improving hemiparetic upper limb motor functionality and modulating cortical excitation/inhibition in patients with stroke.

Hypothesis to be tested: We hypothesize that low intensity priming iTBS can maximize the induction of therapeutically beneficial metaplasticity, and that this will be reflected in enhanced cortical excitation and reduced cortical inhibition, thereby enabling superior upper limb motor recovery in patients with stroke.

Design and subjects: A randomized controlled trial involving 108 patients with chronic stroke.

Study instruments: Transcranial magnetic stimulation (TMS) and electroencephalography (EEG).

Interventions: Participants will be randomly assigned into one of the following four groups: (1) low intensity priming iTBS (55% resting motor threshold [RMT] continuous theta burst stimulation [cTBS]+70% RMT iTBS); (2) conventional intensity priming iTBS (70% RMT cTBS+70% RMT iTBS); (3) nonpriming iTBS (sham cTBS+70% RMT iTBS); and (4) sham stimulation (sham cTBS+sham iTBS). All participants will receive 60-minute standard motor training after completion of the stimulation program. The intervention will last four weeks, with three sessions per week.

Main outcome measures: Upper limb motor tests and levels of cortical excitation/inhibition measured by TMS-evoked EEG potentials.

Data analysis: Analysis of variance (ANOVA). Expected results: The low intensity priming iTBS protocol will be the most efficacious protocol for enhancing cortical excitation and reducing cortical inhibition in post-stroke patients and will thereby produce superior outcomes with regard to upper limb motor functionality.

ELIGIBILITY:
Inclusion Criteria

1. Unilateral upper limb motor dysfunction caused by ischemic stroke, with stroke onset≥6 months. Diagnosis will be verified using discharge summary and radiological reports issued by Hospital Authority. Qualifying participants will undergo structural magnetic resonance imaging (MRI) at the University Research Facility in Behavioral and Systems Neuroscience (UBSN) at PolyU to further confirm their lesion location in the period of experimental participation.
2. Age between 18 and 80 years.
3. Residual upper limb functions between levels 2-6 in the FTHUE, indicating moderately-to-severely impaired upper limb motor functions.
4. Capable of providing informed written consent. Exclusion Criteria

Patients who meet any of the following criteria will be excluded:

1. any contraindications to TMS (screened by the safety checklist by Rossi(33)) and/or MRI (screened by the MRI safety checklist offered by UBSN [see supplement]).
2. Diagnosed with any concomitant neurological disease other than stroke.
3. signs of cognitive impairment, with a Montreal cognitive assessment score<21/22 out of 30 (34).
4. Severe spasticity in the hemiparetic upper limb muscles, with a Modified Ashworth score > 2 (35).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
The Fugl-Meyer Assessment-Upper Extremity Scores | Baseline
  The Fugl-Meyer Assessment-Upper Extremity Scores (FMA-UE) is the gold standard for evaluating poststroke upper limb motor control. This assessment is used to determine the movement, coordination, and reflex actions of the hemiplegic upper limb
The Fugl-Meyer Assessment-Upper Extremity Scores | At 3 weeks
  The Fugl-Meyer Assessment-Upper Extremity Scores (FMA-UE) is the gold standard for evaluating poststroke upper limb motor control. This assessment is used to determine the movement, coordination, and reflex actions of the hemiplegic upper limb
The Fugl-Meyer Assessment-Upper Extremity Scores | At one-month
  The Fugl-Meyer Assessment-Upper Extremity Scores (FMA-UE) is the gold standard for evaluating poststroke upper limb motor control. This assessment is used to determine the movement, coordination, and reflex actions of the hemiplegic upper limb

SECONDARY OUTCOMES:
P30 amplitude in the TMS-evoked potential | Baseline
  TMS-evoked potential is a time-locked signal elicited by single TMS pulses delivered to the cortex. P30 means the positive peak appeared at 30 ms after stimulation. The amplitude of P30 is correlated with cortical excitability mediated by excitatory interneurons.
P30 amplitude in the TMS-evoked potential | At 3 weeks
  TMS-evoked potential is a time-locked signal elicited by single TMS pulses delivered to the cortex. P30 means the positive peak appeared at 30 ms after stimulation. The amplitude of P30 is correlated with cortical excitability mediated by excitatory interneurons.
P30 amplitude in the TMS-evoked potential | At one-month
  TMS-evoked potential is a time-locked signal elicited by single TMS pulses delivered to the cortex. P30 means the positive peak appeared at 30 ms after stimulation. The amplitude of P30 is correlated with cortical excitability mediated by excitatory interneurons.

CONTACTS AND LOCATIONS:
Locations (1):
- Jack Jiaqi Zhang, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided